CLINICAL TRIAL: NCT02636595
Title: A Single-Arm, Open-Label Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Adults With Chronic Hepatitis C Virus Genotype 4, 5, or 6 Infection (ENDURANCE-4)
Brief Title: The Efficacy and Safety of ABT-493/ABT-530 in Adults With Chronic Hepatitis C Virus Genotype 4, 5, or 6 Infection (ENDURANCE-4)
Acronym: ENDURANCE-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-583; 2015-002349-80 (EudraCT Number)
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Genotype 4; Hepatitis C; Chronic Hepatitis C; Hepatitis C Genotype 6; Hepatitis C Genotype 5
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-493/ABT-530 (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks.
  Interventions: Drug: ABT-493/ABT-530

INTERVENTIONS:
Drug: ABT-493/ABT-530 — Tablet; ABT-493 coformulated with ABT-530
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; MAVYRET

SUMMARY:
The purpose of this study is to evaluate the effect of response to treatment by evaluating the percentage of subjects achieving a 12-week sustained virologic response (SVR12) after 12 weeks of treatment with ABT-493/ABT-530 and to evaluate the safety of the regimen in participants with chronic hepatitis C virus (HCV) genotype (GT) 4, 5, or 6 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Screening laboratory result indicating hepatitis C virus (HCV) genotype (GT) 4, 5, or 6 infection.
2. Chronic HCV infection.
3. HCV treatment-naïve or treatment experienced (interferon [IFN] or pegylated interferon [pegIFN] with or without ribavirin [RBV]; sofosbuvir [SOF] plus RBV with or without pegIFN).
4. Non-cirrhotic participants.

Exclusion Criteria:

1. History of severe, life-threatening or other significant sensitivity to any excipient of the study drugs.
2. Female who is pregnant, planning to become pregnant during the study, or breastfeeding; or male whose partner is pregnant or planning to become pregnant during the study.
3. Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
4. Positive test result at Screening for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab).
5. Co-infection with more than one HCV genotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Background] Asselah T, Kowdley KV, Zadeikis N, Wang S, Hassanein T, Horsmans Y, Colombo M, Calinas F, Aguilar H, de Ledinghen V, Mantry PS, Hezode C, Marinho RT, Agarwal K, Nevens F, Elkhashab M, Kort J, Liu R, Ng TI, Krishnan P, Lin CW, Mensa FJ. Efficacy of Glecaprevir/Pibrentasvir for 8 or 12 Weeks in Patients With Hepatitis C Virus Genotype 2, 4, 5, or 6 Infection Without Cirrhosis. Clin Gastroenterol Hepatol. 2018 Mar;16(3):417-426. doi: 10.1016/j.cgh.2017.09.027. Epub 2017 Sep 22. PMID 28951228
- [Derived] Brown A, Welzel TM, Conway B, Negro F, Brau N, Grebely J, Puoti M, Aghemo A, Kleine H, Pugatch D, Mensa FJ, Chen YJ, Lei Y, Lawitz E, Asselah T. Adherence to pan-genotypic glecaprevir/pibrentasvir and efficacy in HCV-infected patients: A pooled analysis of clinical trials. Liver Int. 2020 Apr;40(4):778-786. doi: 10.1111/liv.14266. Epub 2019 Oct 18. PMID 31568620
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Gane E, Poordad F, Zadeikis N, Valdes J, Lin CW, Liu W, Asatryan A, Wang S, Stedman C, Greenbloom S, Nguyen T, Elkhashab M, Worns MA, Tran A, Mulkay JP, Setze C, Yu Y, Pilot-Matias T, Porcalla A, Mensa FJ. Safety and Pharmacokinetics of Glecaprevir/Pibrentasvir in Adults With Chronic Genotype 1-6 Hepatitis C Virus Infections and Compensated Liver Disease. Clin Infect Dis. 2019 Oct 30;69(10):1657-1664. doi: 10.1093/cid/ciz022. PMID 30923816
- [Derived] Foster GR, Dore GJ, Wang S, Grebely J, Sherman KE, Baumgarten A, Conway B, Jackson D, Asselah T, Gschwantler M, Tomasiewicz K, Aguilar H, Asatryan A, Hu Y, Mensa FJ. Glecaprevir/pibrentasvir in patients with chronic HCV and recent drug use: An integrated analysis of 7 phase III studies. Drug Alcohol Depend. 2019 Jan 1;194:487-494. doi: 10.1016/j.drugalcdep.2018.11.007. Epub 2018 Nov 24. PMID 30529905
- [Derived] Flamm S, Reddy KR, Zadeikis N, Hassanein T, Bacon BR, Maieron A, Zeuzem S, Bourliere M, Calleja JL, Kosloski MP, Oberoi RK, Lin CW, Yu Y, Lovell S, Semizarov D, Mensa FJ. Efficacy and Pharmacokinetics of Glecaprevir and Pibrentasvir With Concurrent Use of Acid-Reducing Agents in Patients With Chronic HCV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):527-535.e6. doi: 10.1016/j.cgh.2018.07.003. Epub 2018 Sep 10. PMID 30012435
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 35-day screening period.
Period: Overall Study
Arm/Group | ABT-493/ABT-530
Started | 121
Completed | 119
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.66 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 77

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat (ITT) population: all participants who received at least 1 dose of study drug; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 121
percentage of participants | 99.2 [97.6 to 100]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline HCV RNA during treatment; confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment, or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Treatment weeks 1, 2, 4, 8, and 12 (end of treatment) or premature discontinuation from treatment
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 121
percentage of participants | 0 [0.0 to 3.1]

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment, excluding reinfection.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 118
percentage of participants | 0 [0.0 to 3.2]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE with an onset date after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ABT-493/ABT-530
Serious Adverse Events (participants affected / at risk) | 1/121
Other Adverse Events (participants affected / at risk) | 59/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-493/ABT-530 (N=121)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-493/ABT-530 (N=121)
DIARRHOEA (Gastrointestinal disorders) | 8
NAUSEA (Gastrointestinal disorders) | 12
ASTHENIA (General disorders) | 11
FATIGUE (General disorders) | 21
HEADACHE (Nervous system disorders) | 25
PRURITUS (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.